CLINICAL TRIAL: NCT06378827
Title: The Effect of Intraoperative Dexmedetomidine on Renal Function After Coronary Artery Bypass Graft Surgery
Brief Title: Intraoperative Dexmedetomidine and Coronary Artery Bypass Graft Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Ranko Zdravkovic, Principal Investigator, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 418-1/2
Record Dates: First submitted 2024-04-13; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients from the experimental group will receive a continuous infusion of dexmedetomidine at a dose of 0.5 µg/kg/h, until the end of the operation.
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator): Patients in the control group will receive the same volume of saline solution.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine solution will be prepared by diluting one ampoule of dexmedetomidine (200µg/2ml) with 48 ml of saline solution to obtain a dexmedetomidine solution of 4µg/ml. Patients from the experimental group will receive a continuous infusion of dexmedetomidine at a dose of 0.5 µg/kg/h, until the end of the operation.

SUMMARY:
This is a prospective randomized clinical trial designed to determine the effect of intraoperative dexmedetomidine administration on renal function after coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
This study will include patients admitted to the Clinic for Cardiovascular Surgery of the Institute of Cardiovascular Diseases of Vojvodina, planned for elective coronary artery bypass graft surgery (CABG). Basic demographic and anthropometric data (gender, age, height, weight, and body mass index) and data on comorbidities, therapy, and allergies will be recorded. The day before surgery, all patients will undergo transthoracic echocardiography, on the basis of which the ejection fraction of the left ventricle will be determined and recorded. After the entire examination, the New York Heart Association (NYHA) class, American Society of Anaesthesiologists physical status (ASA score), and Estimate risk of in-hospital death after cardiac surgery score (EuroSCORE II) will be determined. The method and purpose of the research will be explained to all patients, after which informed consent for participation in the research will be obtained.

The patients will be divided into two groups (experimental and control) using the randomization method. All patients will have blood drawn for laboratory and biochemical analyses the morning before surgery: urea, creatinine, cystatin C, IL-6, hemoglobin, leukocytes, platelets, glycemia, aspartate aminotransferase (AST), alanine transaminase (ALT), lactate dehydrogenase (LDH), direct and total bilirubin, fibrinogen, CRP, CK-MB, hS troponin I, electrolytes (Na+ and K+), and lactates. With the help of the Cockcroft-Gault formula, the estimated glomerular filtration rate (eGFR) and creatinine clearance (CCr) will be determined. The values of all these analyses will be defined as basal values.

The anesthetic and surgical protocol, as well as the postoperative treatment, will be standardized. Half an hour before arriving in the operating room, patients will receive about 0.05 mg/kg of midazolam per os as premedication. Upon arrival in the operating room, electrodes for continuous monitoring of the electrocardiogram (ECG), electrodes for assessing the depth of anesthesia, and pulse oximetry for monitoring pulse saturation (SpO2) will be attached to all patients. Anesthetist nurses will place a peripheral venous cannula, usually in one of the veins of the right arm, through which infusion solutions will be applied in the perioperative period and if necessary, transfusions of autologous blood, resuspended erythrocytes, platelets, and fresh frozen plasma. The anesthesiologist will place the arterial cannula, mostly in the left radial artery, for continuous monitoring of arterial blood pressure values. After adequate preoxygenation (8 l/min, 3 min) via a ventilation mask, the intravenous anesthesia will be administered with a combination of the benzodiazepine midazolam (about 0.05 mg/kg), the opioid analgesic sufentanil (about 0.15 µg/kg), intravenous anesthetic propofol (about 1 mg/kg), and the neuromuscular relaxant rocuronium bromide (about 0.8 mg/kg). After endotracheal intubation, patients will be on mechanical lung ventilation (MLV) - volume-controlled ventilation mode with a tidal volume of 6-8 ml/kg of ideal body weight, a respiratory rate of 12/min, FiO2 of 0.5, a positive end-expiratory pressure (PEEP) of 5 cmH2O, and an inspiratory ratio to expirium - I:E 1:2. The flow of fresh gases at the MLV in all patients will be 3 l/min. Correction of MLV parameters will be done based on partial pressures of oxygen (PaO2) and carbon dioxide (PaCO2) in arterial blood, with the aim of maintaining PaO2 >100 mmHg and PaCO2 35-45 mmHg. A three-lumen central venous catheter (CVC) will be placed mainly in the right interior jugular vein. All patients will be placed with a urinary catheter to monitor hourly diuresis as well as a nasopharyngeal probe to monitor nasopharyngeal temperature.

Dexmedetomidine solution will be prepared by diluting one ampoule of dexmedetomidine (200µg/2ml) with 48 ml of saline solution to obtain a dexmedetomidine solution of 4µg/ml. Patients from the experimental group will receive a continuous infusion of dexmedetomidine at a dose of 0.5 µg/kg/h, until the end of the operation. Patients in the control group will receive the same volume of saline solution.

Anesthesia will be maintained with the inhaled anesthetic sevoflurane, with target depth of anesthesia values between 40 and 60, as measured by entropy. A continuous intravenous infusion of sufentanil (0.5-1 µg/kg/h) will be used for intraoperative analgesia. Neuromuscular relaxation will be maintained by intermittent bolus doses of rocuronium bromide (on average, about 0.4 mg/kg/h). All patients will receive an intravenous antibiotic (Ceftriaxone 1g) half an hour before the surgical incision, and in cases of allergy to cephalosporins, Vancomycin 500 mg. All patients are prescribed tranexamic acid according to the protocol.

All operations will be performed through a medial sternotomy approach. To achieve total heparinization, heparin will be prescribed at a dose of 300-400 IU/kg. After 5 minutes from the administration of heparin, arterial blood will be drawn to determine the activated coagulation time, i.e, ACT. After reaching the value of ACT >480 s, cardiopulmonary bypass (CPB) will be started. During that period, the inhalation anesthetic will be turned off, and anesthesia will be maintained with a continuous infusion of propofol. During the application of the CBP pump, MLV will be performed with a tidal volume of 2-3 ml/kg of ideal body weight, a respiratory rate of 10/min, an FiO2 of 0.5, and a PEEP of 5 cmH2O. Membrane oxygenators will be used for CPB, which will be "primed" with 1500 ml of Hartmann's solution and 2500 IU of heparin. The flow rate of the CPB non-pulsating pump will be 2-2.4 l/min/m2. The value of mean arterial pressure during CPB will be maintained between 50 and 80 mmHg. Hemoglobin values will be maintained above 8 g/dl, and hematocrit values will be above 0.22. In cases of lower values, resuspended erythrocytes will be prescribed. Crystalloid cardioplegic solution or blood cardioplegia will be used to stop and protect the myocardium. All operations will be performed under conditions of mild hypothermia (33-34°C). It will be recorded whether the heart, after removing the aortic clamp, worked spontaneously, whether it was defibrillated with an internal defibrillator, or whether a temporary pacemaker was applied. To reverse the effect of heparin, after the completion of CPB and removal of the cannula for CPB, protamine sulfate will be prescribed at a dose of 1 mg per 100 IU of heparin.

During the operation, the anesthesiologist will record the values of systolic and diastolic arterial blood pressure and heart rate every 5 minutes, the values of central venous pressure, SpO2, and depth of anesthesia every 15 minutes, as well as hourly diuresis in the anesthesia chart. The presence of significant arterial hypotension (mean arterial pressure < 65 mmHg or < 50 mmHg during CPB) lasting at least 5 min will be recorded, and whether it lasted 5-15, 15-30 or longer than 30 min will be recorded. The length of application of the aortic clamp, the length of application of the CPB pump, and the length of the operation will be recorded. The total doses of propofol (mg), sufentanil (µg), and the volume of sevoflurane (ml) administered during the operation will be recorded, as well as the total volume of Hartmann's solution, cardioplegia solution, and eventual transfusion of autologous blood, resuspended erythrocytes, platelets, and fresh frozen plasma. It will be recorded whether the patient was prescribed antihypertensives, sympathomimetics, parasympatholytics, inotropics, and vasopressor support, in what doses, and for what period of time if a continuous infusion was used.

After surgery, the patients will be sedated with a continuous infusion of propofol (about 2 mg/kg/h) and on MLV and will be transferred to the ICU, where, after meeting the criteria necessary for separation from MLV, they will be extubated. Continuous monitoring (ECG, invasive arterial pressure, central venous pressure, SpO2, hourly diuresis, body temperature, arterial blood gas analysis) continues during the stay of patients in the intensive care unit (ICU) and in the semi-intensive care unit. On the first three days (the day of surgery and the first two postoperative days), the presence of mean arterial pressure < 65 mmHg will be recorded, and it will be noted whether it lasted less than 1 hour, 1-3 hours, 3-6 hours, or more than 6 hours. The intake of crystalloid solutions, resuspended erythrocytes, fresh frozen plasma, and platelets will be monitored and recorded. Daily diuresis, daily blood loss, the amount of prescribed diuretics during 24 hours, as well as the use of inotropes, will be recorded. During the first three days, the presence of oliguria (<0.5 ml/kg) will be recorded and noted, whether it lasted 6-12 hours or longer than 12 hours, the presence of severe oliguria (<0.3 ml/kg) lasting longer than 24 hours, or the presence of anuria lasting longer than 12 hours.

On the first postoperative day, all laboratory and biochemical analyses that were performed preoperatively will be repeated (urea, creatinine, cystatin C, IL-6, hemoglobin, leukocytes, platelets, glycemia, AST, ALT, LDH, direct to total bilirubin, fibrinogen, CRP, CK-MB, hS troponin I, Na+, K+ and lactates). On the second postoperative day, serum cystatin C, creatinine, Na+, K+ and lactate analyses will be repeated. Creatinine values will be determined on the third and fifth postoperative day. Based on each new creatinine value, eGFR and CCr will be determined.

For all patients, the length of postoperative MLV (in hours), the length of stay in the ICU (in days), the length of hospitalization after surgery (in days), and possibly death will be recorded.

The primary objective of the study will be to monitor and compare, between groups, indicators of renal function (serum creatinine, cystatin C, diuresis, eGFR, and CCr). The changes of all these values in relation to the basal values will be monitored, in order to determine when the greatest changes in the values of the indicators of renal function occur. Of particular importance will be the correlation between serum cystatin C and creatinine values. During the first three days, daily diuresis, the volume of prescribed liquids, the administration and doses of diuretics, and the values of Na+, K+, and lactate will be monitored and compared. The frequency of the occurrence of acute kidney injury (AKI) will be monitored. The diagnosis of AKI will be based on the criteria of the KDIGO guide.

The change of inflammatory markers (IL-6, CRP, leukocytes, fibrinogen) in relation to basal values is also one of the primary goals of the research. Inflammatory markers will be checked on the first postoperative day, when the inflammatory response is most pronounced. A correlation will be made between IL-6 and other inflammatory markers that are in routine clinical use (CRP, leukocytes, and fibrinogen) in order to determine which inflammatory marker correlates best with IL-6. A correlation between IL-6 values and serum creatinine and cystatin C values will also be performed, in order to determine whether impairment of renal function is related to the intensity of the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery bypass graft surgery
* Age over 18 years
* ASA score 3 or 4
* Voluntary consent of the patient to participate in the research

Exclusion Criteria:

* Emergency coronary artery bypass graft surgery
* Chronic renal failure with eGFR <60 ml/min/1.73m2
* Left ventricular ejection fraction <30%
* 2nd or 3rd degree atrioventricular block
* Use of nephrotoxic agents such as aminoglycoside antibiotics or contrast agents within the last 48 hours
* Previous heart surgery or kidney surgery
* Allergy to dexmedetomidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Indicator of renal function | 5 days
  The primary objective of the study will be to monitor serum creatinine (µmol/L) and compare between groups. The changes of all these values in relation to the basal values will be monitored in order to determine when the greatest changes in the serum creatinine values occur.
An early biomarker of kidney injury | 2 days
  The primary objective of the study will be to monitor serum cystatin C (mg/L) and compare between groups. The changes of all these values in relation to the basal values will be monitored in order to determine when the greatest changes in the serum cystatin C values occur.
The change of inflammatory markers | 24 hours
  The change of inflammatory marker IL-6 (pg/mL) in relation to basal values is also one of the primary goals of the research. IL-6 will be checked on the first postoperative day, when the inflammatory response is most pronounced.

SECONDARY OUTCOMES:
Length of postoperative mechanical ventilation | 24 hours
  The length of postoperative mechanical ventilation (hours) will be compared.
Length of stay in the intensive care unit | 3 days
  The length of stay in the intensive care unit will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- University of Novi Sad, Faculty of Medicine, Novi Sad, Serbia

REFERENCES:
- [Derived] Zdravkovic R, Vickovic S, Preveden M, Drobnjak V, Lukic-Sarkanovic M, Miljevic IB, Tatic M, Tubic T, Videnovic N, Mladenovic N, Komazec N, Dracina N, Jerkovic M, Djokovic A, Jakovljevic A, Kostic A, Mehmedi E, Redzek A. Effect of Continuous Intraoperative Dexmedetomidine on Interleukin-6 and Other Inflammatory Markers After Coronary Artery Bypass Graft Surgery: A Randomized Controlled Trial. Medicina (Kaunas). 2025 Apr 24;61(5):787. doi: 10.3390/medicina61050787. PMID 40428745